CLINICAL TRIAL: NCT01498822
Title: A Multi-Center, Open-label, Randomized Study to Evaluate the Long Term Effectiveness of Levetiracetam as Monotherapy in Comparison With Oxcarbazepine in Subjects With Newly or Recently Diagnosed Partial Epilepsy
Brief Title: Levetiracetam Versus Oxcarbazepine as Monotherapy to Evaluate Efficacy and Safety in Subjects With Newly or Recently Diagnosed Partial Epilepsy
Acronym: OPTIMAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea UCB Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N01367; 2014-002713-32 (EudraCT Number)
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Results first posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-07

CONDITIONS: Epilepsy
Keywords: Levetiracetam; Oxcarbazepine; treatment failure; partial epilepsy
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial | interventions — Levetiracetam; Oxcarbazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levetiracetam (Experimental): Levetiracetam twice a day treatment group
  Interventions: Drug: Levetiracetam
- Oxcarbazepine (Active Comparator): Oxcarbazepine twice a day treatment group
  Interventions: Drug: Oxcarbazepine

INTERVENTIONS:
Drug: Levetiracetam — 250 mg and 500 mg Levetiracetam tablet, 1000 mg-3000 mg/day, maximum 50 weeks including initial up titration of 500 mg/day for 2 weeks
  Arms: Levetiracetam
Drug: Oxcarbazepine — 150 mg and 300 mg Oxcarbazepine tablet, 900 mg-2400 mg/day, maximum 50 weeks including 2 weeks of up titration (300 mg/day 1week then 600 mg/day 1 week)
  Arms: Oxcarbazepine

SUMMARY:
To evaluate the long term effectiveness of Levetiracetam (LEV) monotherapy on Treatment Failure Rate in subjects with newly diagnosed partial onset seizures with or without secondary generalized seizures, compared to Oxcarbazepine (OXC) monotherapy over 50 weeks from the first dose

DETAILED DESCRIPTION:
The study duration consists of the following periods:

* Baseline period of one week: Week -1
* Titration period of two weeks: Week 0 to Week 1
* Treatment period of 48 weeks: Week 2 to Week 50

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects from 16 to 80 years, inclusive. Vulnerable subjects (e.g., under 20 years or subject with learning disability but judged to be capable to understand) may only be included where legally permitted and ethically accepted
* Subjects with newly or recently diagnosed epilepsy having experienced unprovoked partial seizures (IA, IB, IC with clear focal origin), that are classifiable according to the International Classification of Epileptic seizure (1981). Undiscriminated subjects between IC and IIE could be included
* Subjects with at least 2 unprovoked seizures separated by a minimum of 48 hours in the year preceding randomization out of which at least 1 unprovoked seizure in the 6 months preceding randomization
* Subjects with documented evidence of EEG and brain MRI or CT scan in medical records which were performed within 1 year prior to Visit 1 (V1)
* Subjects have no treatment with anti-epileptic drugs in the 6 months preceding this study. The treatment for acute seizure control is acceptable with a maximum of 2 weeks duration and if the treatment was stopped at least 1 week before V1. For Phenobarbital and Phenobarbital derivatives, a minimum of 4 weeks wash-out is requested before V1

Exclusion Criteria:

* Subject has a current or previous diagnosis of pseudoseizures, conversion disorders, or other non-epileptic ictal events which could be confused with seizures
* Subject taking 1 or more of the following medications on a regular basis within 28 days prior to Visit 1: neuroleptics, monoamine oxidase (MAO) inhibitors and narcotic analgesics
* Subject taking any immunosuppressant within 28 days prior to Visit 1
* Subject has a history of suicide attempt, has received professional counseling for suicidal ideation, or is currently experiencing active suicidal ideation
* Subject has a seizure disorder characterized primarily by isolated auras (ie, simple partial seizures without observable motor signs)
* Subject suffering from seizures other than partial (IA, IB, IC, with clear focal origin) seizures
* Subject has a history of status epilepticus within last 3-month period prior to Visit 1
* Subject has seizures that are uncountable due to clustering (ie, an episode lasting less than 30 minutes in which several seizures occur with such frequency that the initiation and completion of each individual seizure cannot be distinguished) during the 12-week period prior to Visit 1 and/or during the Screening Period
* Body weight is lower than 40 kg (< 40 kg)

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2011-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (23):
- South Korea (23):
  - 05, Busan
  - 10, Busan
  - 16, Busan
  - 06, Daejeon
  - 18, Daejeon
  - 23, Gangwon-Do
  - 08, Goyang-si
  - 09, Goyang-si
  - 07, Gwangju
  - 22, Junggu
  - 14, Seongnam-si
  - 01, Seoul
  - 02, Seoul
  - 03, Seoul
  - 04, Seoul
  - 11, Seoul
  - 12, Seoul
  - 13, Seoul
  - 15, Seoul
  - 17, Seoul
  - 20, Seoul
  - 21, Seoul
  - 19, Ulsan

REFERENCES:
- [Derived] Kim JH, Lee SK, Loesch C, Namgoong K, Lee HW, Hong SB; Korean N01367 Study Group. Comparison of levetiracetam and oxcarbazepine monotherapy among Korean patients with newly diagnosed focal epilepsy: A long-term, randomized, open-label trial. Epilepsia. 2017 Apr;58(4):e70-e74. doi: 10.1111/epi.13707. PMID 28395124
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll subjects in June 2011. A total of 27 investigators enrolled 353 subjects at 23 sites in Korea.
Pre-assignment Details: Participant Flow refers to the Randomized Set, consisting of all subjects who were randomized in this study.
Groups:
- Oxcarbazepine: Oxcarbazepine twice a day treatment Group
  150 mg and 300 mg Oxcarbazepine tablet, 900 mg-2400 mg/day, maximum 50 weeks including 2 weeks of up titration (300 mg/day 1 week then 600 mg/day 1 week)
Period: Overall Study
Arm/Group | Levetiracetam | Oxcarbazepine
Started | 175 | 178
Completed | 121 | 122
Not Completed | 54 | 56
Not completed — Protocol Violation | 8 | 4
Not completed — Other Reason | 5 | 2
Not completed — Lack of Efficacy | 7 | 2
Not completed — AE, non-serious non-fatal | 8 | 17
Not completed — SAE, non-fatal | 2 | 2
Not completed — Adverse Event, serious fatal | 1 | 1
Not completed — Withdrawal by Subject | 15 | 25
Not completed — Lost to Follow-up | 8 | 3

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Randomized Set, consisting of all subjects who were randomized in this study.
Arm/Group | Levetiracetam | Oxcarbazepine | Total Title
Number analyzed (Participants) | 175 | 178 | 353
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 13 | 27
  Between 18 and 65 years | 145 | 143 | 288
  >=65 years | 16 | 22 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (16.7) | 42.7 (17.3) | 41.1 (17.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 79 | 163
  Male | 91 | 99 | 190
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 174 | 178 | 352
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With a Treatment Failure
Description: Treatment failure is defined as (1) Dropout due to related intolerable adverse event, lack of efficacy or need for addition of another Antiepileptic Drug (AED), or (2) need of a 1-step down-Titration, within 50 weeks from the first dose of study medication.
Time Frame: Week 0 (First Dose) to Week 50
Population: Per Protocol Set (PPS) consisted of all subjects who received at least 1 (partial) dose of study mediaction, returned at least 1 post-Baseline seizure diary and had no important protocol deviations. Subjects who discontinued the study before Week 50 for any reason other than treatment failure were excluded from the PPS.
Measure: Number; unit: percentage of subjects
Groups:
- Per Protocol Set (LEV Treated Subjects): 250 mg and 500 mg Levetiracetam tablet, 1000 mg-3000 mg/day, maximum 50 weeks including initial up titration of 500 mg/day for 2 weeks
- Per Protocol Set (OXC Treated Subjects): 150 mg and 300 mg Oxcarbazepine tablet, 900 mg-2400 mg/day, maximum 50 weeks including 2 weeks of up titration (300 mg/day 1 week then 600 mg/day 1 week)
Arm/Group | Per Protocol Set (LEV Treated Subjects) | Per Protocol Set (OXC Treated Subjects)
Number analyzed (Participants) | 118 | 128
percentage of subjects | 12.7 | 23.4
Statistical Analysis 1: Comparison: Per Protocol Set (LEV Treated Subjects) vs Per Protocol Set (OXC Treated Subjects); Test type: Non-Inferiority or Equivalence — The primary analysis of this study aimed to demonstrate that LEV was noninferior to OXC with respect to the treatment failure rate in the Per Protocol Set. The noninferiority margin was 15 %; Wald methodology; Absolut difference = -10.7, 95% CI 2-sided [-20.2 to -1.2] — Absolute difference in treatment failure rates of LEV versus OXC is defined as "Treatment Failure Rate LEV" minus "Treatment Failure Rate OXC"

2. Secondary Outcome: Time to the First Seizure Defined as the Time From the First Dose of Medication to the Occurrence of the First Seizure During the 48 Weeks Treatment Period
Time Frame: From Week 2 to Week 50 (During Treatment Period )
Population: The Full Analysis Set (FAS) consisted of all subjects who received at least 1 (partial) dose of study mediaction and returned at least 1 post-Baseline seizure diary.
  A randomized subject was only excluded from the FAS when there was clear evidence that the subject did not take any study medication.
Measure: Median (Full Range); unit: months
Groups:
- Full Analysis Set (LEV Treated Subjects): 250 mg and 500 mg Levetiracetam tablet, 1000 mg-3000 mg/day, maximum 50 weeks including initial up titration of 500 mg/day for 2 weeks
- Full Analysis Set (OXC Treated Subjects): 150 mg and 300 mg Oxcarbazepine tablet, 900 mg-2400 mg/day, maximum 50 weeks including 2 weeks of up titration (300 mg/day 1 week then 600 mg/day 1 week)
Arm/Group | Full Analysis Set (LEV Treated Subjects) | Full Analysis Set (OXC Treated Subjects)
Number analyzed (Participants) | 173 | 171
months | 7.556 [NA to NA] — Dispersion measures for this statistic were not part of the analysis (or it's specification). | NA [NA to NA] — Kaplan-Meier estimation of percentage of event-free subjects does not fall to or below 50 %, therefore no median time to event could be estimated for the OXC group.

3. Secondary Outcome: Percentage of Subjects Who Achieved Seizure Freedom for 24 Consecutive Weeks During the 48 Weeks Treatment Period at Any Time
Description: 24-week Seizure Freedom (rate) defined as the number and percentage of subjects who achieved seizure freedom for 24 consecutive weeks during the Treatment Period at any time
Time Frame: From Week 2 to Week 50 (During Treatment Period )
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Full Analysis Set (LEV Treated Subjects) | Full Analysis Set (OXC Treated Subjects)
Number analyzed (Participants) | 173 | 171
percentage of subjects | 53.8 | 58.5

4. Secondary Outcome: Percentage of Subjects Who Achieved Seizure Freedom During the 48 Weeks Treatment Period
Description: 48-week Seizure Freedom (rate) defined as the number and percentage of subjects who achieved seizure freedom during the Treatment Period
Time Frame: From Week 2 to Week 50 (During Treatment Period )
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Full Analysis Set (LEV Treated Subjects) | Full Analysis Set (OXC Treated Subjects)
Number analyzed (Participants) | 173 | 171
percentage of subjects | 34.7 | 40.9

ADVERSE EVENTS:
Time Frame: Adverse Events were collected up to 57 Weeks from Visit 1 (Week -1) to the end of the post-treatment period (down-titration visit, safety follow-up visit).
Description: Adverse Events refer to the Safety Set (SS). SS consisted of all subjects who were randomized and received at least 1 (partial) dose of study medication.
Arm/Group | Levetiracetam | Oxcarbazepine
Serious Adverse Events (participants affected / at risk) | 15/173 | 15/174
Other Adverse Events (participants affected / at risk) | 67/173 | 93/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=173) | Oxcarbazepine (N=174)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 4 (4) | 5 (5)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abortion induced (Surgical and medical procedures) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=173) | Oxcarbazepine (N=174)
Nasopharyngitis (Infections and infestations) | 14 (15) | 19 (21)
Dizziness (Nervous system disorders) | 25 (30) | 50 (70)
Headache (Nervous system disorders) | 25 (29) | 36 (53)
Somnolence (Nervous system disorders) | 22 (30) | 24 (30)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 13 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days